CLINICAL TRIAL: NCT02840448
Title: Impact of Elastin Mediated Vascular Stiffness on End Organs
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160144; 16-H-0144
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-12-17

CONDITIONS: Williams Syndrome; Supravalvular Aortic Stenosis; Cardiovascular Disease
Keywords: Williams Syndrome; Blood Flow; Brain; Arterial Stiffness; Natural History; Variation in WS Genes
MeSH Terms: conditions — Williams Syndrome; Aortic Stenosis, Supravalvular; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Subjects with WS/SVAS/WS gene region variation
- Controls: Healthy volunteers

SUMMARY:
Background:

People with Williams Syndrome (WS) and supravalvular aortic stenosis (SVAS) have less elasticity in their blood vessels. This is called blood vessel stiffness. Blood vessels may have focal narrowings called stenoses or may just be globally more narrow.

Objectives:

Researchers want to see how blood vessel differences in people with Williams Syndrome and supravalvular aortic stenosis affect organs in the body including the heart, gut, kidneys, and brain.

Eligibility:

People ages 3-85 who have WS or SVAS

Healthy volunteers ages 3-85

Design:

* Participants will have yearly visits for up to 10 years. All participants will be offered the same tests.
* Participants will give consent for the study team to review their medical records. If the participant is a child or an adult with WS, a parent or guardian will give the consent.
* Participants will visit the NIH where they will have a physical exam and medical history. Based on their health history, participants will undergo a series of imaging tests and measures of blood vessel function over the course of 2-4 days. Tests of cognitive abilites will also be performed. Blood will be drawn and an IV may be placed for specific tests.

DETAILED DESCRIPTION:
Elasticity in the aorta buffers the body from damage due to pulsatile blood flow. Data from humans and mice show that with increasing age, vessels lose elasticity and become stiff. Vascular stiffness is associated with progressive cognitive impairment and dementia in aging adults, but little is known about the effects of early-onset/congenital vascular stiffness. Similarly, elastin-mediated arteriopathy in the form of stenosis has the potential to impact additional end organs such as the heart, lungs, gut, skeletal muscle and kidney causing feeding and exercise intolerance, as well hypertension. This study evaluates the impact of elastin arteriopathy and vascular stiffness on end organs.

Following consent, the investigators will work with the subjects and their caregivers to determine which tests are most appropriate for the patient based on their age/capabilities and preferences and may include:

* testing of cognitive and neurobehavioral abilities as well as measures of general health and well being
* undergo non-invasive measurements of vascular stiffness
* undergo brain imaging by MRI
* undergo echocardiogram
* undergo ECG
* undergo 24-hour ambulatory electrocardiogram monitor
* undergo ultrasound imaging and flow studies of various vascular beds and tissues
* undergo CT angiogram of relevant vessels
* undergo non-invasive tissue oxygenation and endothelial functional assessment with near infrared spectroscopy (NIRS) of the limbs and/or head/brain (fNIRS)
* perform a 6 minute walk test
* perform pulmonary function tests
* receive an eye exam and Optical coherence tomography (OCT)
* give blood/urine for relevant laboratories
* evaluate biomechanical properties of skin
* evaluate baseline fitness information using a fitness tracker
* complete medica photography evaluating relevant features of the condition
* receive a dental examination and dental photography

Visits may be conducted in person at the Clinical Center, by telehealth, or with a combination of in person and telehealth, at the discretion of the study team. All telehealth activities will be performed according to HRPP Policy 303 and only testing that can be performed at home (e.g. clinical consultations, neurobehavioral testing, fitness tracking, ambulatory ecg monitoring, and photography) will be selected. The other tests require the individual to be on site at the CC.

Consequently, some participants may have certain consultations at home and other testing on site to limit time in the CC

Additionally, the study will request permission to review the participant's medical records to obtain additional information about general and cardiovascular health. For individuals with supravalvular aortic stenosis (SVAS) or Williams syndrome (WS), the clinical report confirming the individuals diagnosis will be reviewed when available.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will recruit individuals with people with WS, SVAS or other WS region variation conditions (cases) and demographically similar control (unaffected) participants.

Children or adults with WS must:

* be between the ages of 3 and 85
* have a presumed or confirmed diagnosis of WS (genetic testing is not performed in this research study).
* have a parent/guardian available to provide consent and assist in answering medical questions
* not be pregnant

Children or adults with SVAS must:

* be between the ages of 3 and 85
* have clinical features suggestive of SVAS or an SVAS-like condition OR have no clinical features of SVAS or an SVAS-like condition but have genetic testing results that imply affected status (SVAS has decreased penetrance). No genetic testing will be done as part of this protocol.
* have a parent/guardian available to provide consent and assist in answering medical questions if they are a minor (not applicable to adults)

Children or adults with WS region gene changes:

* be between the ages of 3 and 85
* have clinical or research genetic testing that reports gene variation in a non-ELN gene in the WS region.
* have a parent/guardian available to provide consent and assist in answering medical questions if they are a minor or if they have cognitive impairment that would impede their ability to consent on their own behalf.

Children or adults participating in the study as part of control group must:

* be between the ages of 3 and 85
* not have clinical features or genetic profile suggestive of WS, SVAS or an SVAS-like condition. No genetic testing will be performed in this research study.
* have a parent/guardian available to provide consent and assist in answering medical questions if they are a minor (not applicable to adults)

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical along with matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
By testing both WS and SVAS and WS gene region variation subgroups, we can investigate both the effect of elastin insufficiency mediated vascular disease on end organ function and look for a synergistic effect of the larger gene deletion on elas... | ongoing
  Pilot studies aimed at identifying differences between the WS/SVAS/WS gene region variation population and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Boehm, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Washington University School of medicine, St Louis, Missouri

REFERENCES:
- [Background] Pober BR. Williams-Beuren syndrome. N Engl J Med. 2010 Jan 21;362(3):239-52. doi: 10.1056/NEJMra0903074. No abstract available. PMID 20089974
- [Background] Franklin SS. Beyond blood pressure: Arterial stiffness as a new biomarker of cardiovascular disease. J Am Soc Hypertens. 2008 May-Jun;2(3):140-51. doi: 10.1016/j.jash.2007.09.002. PMID 20409896
- [Background] Gorelick PB, Scuteri A, Black SE, Decarli C, Greenberg SM, Iadecola C, Launer LJ, Laurent S, Lopez OL, Nyenhuis D, Petersen RC, Schneider JA, Tzourio C, Arnett DK, Bennett DA, Chui HC, Higashida RT, Lindquist R, Nilsson PM, Roman GC, Sellke FW, Seshadri S; American Heart Association Stroke Council, Council on Epidemiology and Prevention, Council on Cardiovascular Nursing, Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Vascular contributions to cognitive impairment and dementia: a statement for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Sep;42(9):2672-713. doi: 10.1161/STR.0b013e3182299496. Epub 2011 Jul 21. PMID 21778438
- [Derived] Levin MD, Cathey BM, Smith K, Osgood S, Raja N, Fu YP, Kozel BA. Heart Rate Variability Analysis May Identify Individuals With Williams-Beuren Syndrome at Risk of Sudden Death. JACC Clin Electrophysiol. 2023 Mar;9(3):359-370. doi: 10.1016/j.jacep.2022.10.010. Epub 2022 Nov 30. PMID 36752464
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-H-0144.html